CLINICAL TRIAL: NCT07383805
Title: Expression of T Cell Immunoglobulin and Mucin-domain Containing Molecule 3 (Tim-3) on Neutrophils as an Indicator to Assess Disease Activity in Ankylosing Spondylitis Patients
Brief Title: Expression of Tim-3 on Neutrophils in Ankylosing Spondylitis
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Eman Safwat Mohamed, Doctor, Assiut University
Other Study IDs: Tim-AS
Record Dates: First submitted 2026-01-16; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Ankylosing Spondylitis; AS; Tim3
MeSH Terms: conditions — Spondylitis, Ankylosing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. To investigate the expression of Tim-3 on neutrophils in ankylosing spondylitis patients and its correlation with disease activity and inflammatory markers.
2. Association of Tim-3 with sacroiliac MRI findings and the hip inflammatory MRI scoring system (HIMRISS) .

ELIGIBILITY:
Adult patients (>18 years) diagnosed as AS according to 2009 ASAS -Classification criteria (8) Exclusion Criteria:-Age below 18 years old. Patients with other autoimmune diseases. infection (cause increase in inflammatory makers) Any patient with ferromagnetic implants or cardiac pacemaker pregnancy Uncontrolled Hypertension renal failure Chronic liver disease Malignancy Diabetes Mellitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients diagnose as ankylosing spondylitis and healthy controls in Assiut university hospital
Sampling Method: Non-Probability Sample
Enrollment: 81 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
To investigate the expression of Tim-3 on neutrophils in ankylosing spondylitis patients | through study completion, an average of 1 year
  investigate the expression of Tim-3 on neutrophils in ankylosing spondylitis patients and its correlation with disease activity and inflammatory markers

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, University, Egypt

IPD SHARING:
Plan to Share IPD: Undecided